CLINICAL TRIAL: NCT02833428
Title: Acquisition and Analysis of Medullary Trauma Patients Signs, With an Expert Model
Brief Title: Spinal Cord and Artificial Intelligence
Acronym: SKY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SKY
Record Dates: First submitted 2016-07-12; First posted 2016-07-14 (Estimated); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Equipment and Supplies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with acute spinal cord injury (Experimental): The study will be performed on patients with acute spinal cord injury between the cord next to the C2 vertebra and marrow next to the T12 vertebra. This is usually hospitalized patients in an emergency situation, brought by EMS (emergency medical services) and taken care of immediately in the recovery room by intensivists. Patients who accepted to participate to this study will got the installation bedside biomedical equipment for the project (Eclipse Nim, Medtronic®). The aim of this work is to analyze using an artificial intelligence engine (IA, Biomedical equipment (Eclipse Nim, Medtronic®)) the influence of the physiopathological environment (set of parametric data monitoring, imaging, biology etc.) of the traumatized spinal cord on spinal pain.
  Interventions: Device: Biomedical equipment (Eclipse Nim, Medtronic®)

INTERVENTIONS:
Device: Biomedical equipment (Eclipse Nim, Medtronic®) — It is the principal investigator (coordinator investigator moving on the website of the Pitié-Salpêtrière) that will install bedside biomedical equipment for the project (Eclipse Nim, Medtronic®) The term of monitoring will depend of length of stay in the PACU (the post anesthesia care unit) Gaston Cordier and will not exceed 72 hours.
  • Patients will be reviewed at 6 and 12 months for conventional control with establishing a ASIA score (American Spinal Cord Injury Association). Of SEP (Somatosensory evoked potentials) and MEP(Motor Engine Potentials) will be performed in the laboratory at 6 and 12 months (electrophysiology laboratory Pitié-Salpêtrière). They are part of the traditional support in the context of spinal cord trauma.

SUMMARY:
The aim of this study was to analyze using an artificial intelligence engine (IA) the influence of the pathophysiological environment (set parametric monitoring data, imaging, biology etc.) of acute spinal cord trauma on spinal pain. This project seeks to establish the principles of a new approach for studying spinal cord injury patients. It does not meet the usual criteria of clinical trials in so far as it does not test on patients the effect of a therapeutic

DETAILED DESCRIPTION:
Objectives

The objectives are multiple:

1. Analyze clinical situation in the pathophysiology of spinal pain.
2. somatosensory evoked potentials analysis (PES) and motors (PEM) on injuries of the spinal cord in the acute phase.
3. Increasing the mass of data integrated from current standards (volume). The reason is not only an imperative of statistical power as in a conventional test but the probability of specific events characterize this type of pathology and the consequences of their management (monitoring and therapeutic).
4. Identify new predictive parameters and monitoring of spinal pain.

5. Design the tools of computer collection, successful storage formats, adaptations of collection tools: This is validation of the technical solution (i.e. IA).

Expected results

This system will allow to record and analyze a large amount of parameters, largely beyond the human resources. Analysis of these data should allow better understanding of the pathophysiology of acute trauma of the spinal cord which is an essential prerequisite to research new therapies. The realization evoked potentials, ever conducted on this patient in the acute phase should also allow the investigators to better understand the mechanisms of evolution of the SCI (Spinal Cord Injury).

Moreover, this model expert system must allow, through the creation of routines, discovering new predictive parameters and monitoring, improving the management of these patients.

This is a completely open system that can be enriched with new parameters as and above all enriching also as and when the inclusion of new cases. It therefore offers a theoretical field of infinite discovery extremely promising.

ELIGIBILITY:
Inclusion Criteria:

* Patient with acute spinal cord injury between the cord opposite the vertebra C2 and marrow compared to the T12 vertebra.
* neurological lesion classified A, B, C or D according to Frankel classification at the initial examination (Annex 1).
* Patient able to give informed consent

Exclusion Criteria:

There are no exclusion criteria. All patients meeting the inclusion criteria are includable. However, it differs remarkable different situations:

* The clinical neurological assessment of patients may be difficult depending on the context: intubated patients admitted - ventilated multiple trauma.
* Neurological assessment via evoked potentials may be difficult depending on the environment for patient care: need for multiple investigations, resuscitation. Evoked potentials will be installed only after agreement of the healthcare team once the patient is stabilized.
* The patient can refuse to submit to one additional exam is not part of the standard care (i.e. PES / PEM); it will be offered to participate in the study without the completion of this review. It will be in this case a simple use of clinical and laboratory data collected retrospectively anonymized so for scientific purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-01-20 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
Assessment of change of ASIA impairment scale (American Spinal Cord Injury Association) | Day1, 6 months and 1 year
  ASIA impairment scale allows to classify the spinal cord injury according to its level of neurological damage. It is conventionally represented by the most caudal segment having a normal function.
  It allows to appreciate the completeness or incompleteness of the attack. It allows a classification highlighting the severity of the attack by using a five-letter ASIA anomaly scale from A to E.

SECONDARY OUTCOMES:
Assessment of change of Somatosensory Evoked Potentials (SEPs) | Day1, 6 months
  The principal investigator proceeds to the installation of the patient's biomedical material for the project (Nim Eclipse, Medtronic®). The duration of the monitoring will be function the duration of hospitalization in SSPI Gaston Cordier and will not exceed 72 hours. Each night during this period, a non-stimulation range of 6 hours will be provided to allow the included volunteers to sleep.
Assessment of change of Motor Evoked Potentials (PEM) | Day1, 6 months
  The principal investigator proceeds to the installation of the patient's biomedical material for the project (Nim Eclipse, Medtronic®). The duration of the monitoring will be function the duration of hospitalization in SSPI Gaston Cordier and will not exceed 72 hours. Each night during this period, a non-stimulation range of 6 hours will be provided to allow the included volunteers to sleep.

CONTACTS AND LOCATIONS:
Overall Officials: RIOUALLON Guillaume, MD, Principal Investigator — Groupe Hospitalier Paris Saint-Joseph (FRANCE)
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided